CLINICAL TRIAL: NCT04878341
Title: Erector Spinae Plane Block (ESP) Versus Thoracic Epidural Anesthesia in Video-Assisted Thoracoscopic Surgery (VATS) in Pediatric Population; a Randomized, Controlled Study
Acronym: ESP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESP1
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae plane Block (Experimental): After induction of general anesthesia, patients will be positioned in lateral decubitus with surgical site up and the transverse process of T5-T7 vertebrae and Erector Spinae (ES) fascia will be located with a linear ultrasound probe. A 19G or 20G epidural needle (according to age) will be positioned under the ES muscle and a bolus of of 0.3-0.5ml/kg of 0.2% ropivacaine will be administered; after hydrodissection, the catheter will be threaded, followed by an infusion of 0.2mg/kg/hr for the next 48 hours.
  Interventions: Other: Erector Spinae Plane Block
- Thoracic Epidural Anesthesia (Active Comparator): After induction of general anesthesia, patients will be positioned in lateral decubitus with surgical site up and a 19G or 20G epidural needle (according to age) will be positioned at T5-T7 level with cathether placement; a bolus of of 0.3-0.5ml/kg of 0.2% ropivacaine will be administered and followed by an infusion of 0.2mg/kg/hr for the next 48 hours.
  Interventions: Other: Erector Spinae Plane Block

INTERVENTIONS:
Other: Erector Spinae Plane Block — The ESP is fascial plane block performed by injecting local anesthetic between the erector spinae muscle and the transverse process. Its proposed mechanism of action is via blockade of the dorsal and ventral rami of the thoracic spinal nerves and sympathetic fibers.

SUMMARY:
Aim of the study is to investigate the efficacy and safety of continuous ESP block in children under the age of 10 yrs undergoing video-assisted thoracoscopic procedures, compared to Thoracic Epidural Anesthesia (TEA).

DETAILED DESCRIPTION:
Primary outcome:

Post-operative pain assessed by FLACC (Face, Legs, Activity: Cry, Consolability) for children age 1-5 years, and NRS (numerical rating scale) for children age 6-10 years

Secondary outcomes:

* Opioid consumption for 48 hours post-operatively.
* Intraoperative opiod use
* Block failure rate (defined as Heart Rate (HR) increase of more than 20% of baseline at surgical incision)
* Time to extubation after surgery completion After parental consent, children aged 0-10 yrs scheduled for unilateral VATS procedure will be randomized into two groups: Thoracic Epidural Group (TEA) vs Erector Spinae Plane block (ESP).

Children with history of allergy to local anesthetics, systemic coagulopathy, infection at site of puncture, severe renal or liver disease, known rib cage malformations will be excluded from the study.

Anesthesia will be induced at operator's preference; before surgery beginning children will be positioned and either TEA or ESP will be performed. In both cases, a bolus of of 0.3-0.5ml/kg of 0.2% ropivacaine will be administered, followed by an infusion of 0.2mg/kg/hr for the next 48 hours. The time from block placement to incision will be recorded, change in HR before and after incision will be documented, need for intraoperative opiod use, time to first rescue analgesic, and total amount of local anesthetic given at 24 h and 48 h post-operatively will be recorded together with pain measures as specified. Opiods will be prescribed if child presents with FLACC scores > 3 (FLACC score of 0-3 = mild pain, 4-6 = moderate, 7-10 = severe), or VAS >5.

Total opioid consumption will be recorded.

Statistical analysis

Intention to treat analysis will be performed. Quantitative variables will be described as mean and standard deviation (sd) or median and interquartile range (IQR) if not normally distributed (Shapiro-Wilks test) For primary outcome, VAS or FLACC score will be compared with t-test or Mann-Whitney test Opioid consumption will be compared with t-test or Mann-Whitney test Block failure rate will be compared with chi2 test Time to extubation will be compared with log rank test

Sample size With 37 patients for group a power of 80% will be achieved to identify as significant a difference in mean pain score when sd is 1,5 times greater than mean. Alpha error will be 0.05 and a two-sample t-test will be applied.

Randomization A random block centralized randomization list will be generated before study start with Ralloc command in Stata. It will be stratified by center. To avoid allocation concealment the closed envelope method will be used.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Scheduled for Video-Assisted Thoracoscopic Procedure
* Parental consent

Exclusion Criteria:

* Parental refusal
* History of allergy to local anesthetics
* Systemic coagulopathy
* Local infection at puncture site
* Severe renal or liver disease
* Known rib cage malformations

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | First 48 hours after surgery
  Postoperative pain will be assessed by FLACC (Face, Legs, Activity: Cry, Consolability) scale for children aged 1-5 years, and NRS (numerical rating scale) for children aged 6-10 years

SECONDARY OUTCOMES:
Intraoperative opiod use | Surgery duration
  Total amount of intraoperative opiods
Postoperative opiod consumption | First 48 hours after surgery
  Determine if ESP will decrease postoperative opioid consumption compared to Thoracic Epidural Anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Vittore Buzzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swenson Schalkwyk A, Flaherty J, Hess D, Horvath B. Erector spinae catheter for post-thoracotomy pain control in a premature neonate. BMJ Case Rep. 2020 Sep 7;13(9):e234480. doi: 10.1136/bcr-2020-234480. PMID 32900720
- [Background] Gaio-Lima C, Costa CC, Moreira JB, Lemos TS, Trindade HL. Continuous erector spinae plane block for analgesia in pediatric thoracic surgery: A case report. Rev Esp Anestesiol Reanim (Engl Ed). 2018 May;65(5):287-290. doi: 10.1016/j.redar.2017.11.010. Epub 2018 Jan 19. English, Spanish. PMID 29370900
- [Background] De la Cuadra-Fontaine JC, Concha M, Vuletin F, Arancibia H. Continuous Erector Spinae Plane block for thoracic surgery in a pediatric patient. Paediatr Anaesth. 2018 Jan;28(1):74-75. doi: 10.1111/pan.13277. No abstract available. PMID 29226529
- [Background] Patel NV, Glover C, Adler AC. Erector Spinae Plane Catheter for Postoperative Analgesia After Thoracotomy in a Pediatric Patient: A Case Report. A A Pract. 2019 May 1;12(9):299-301. doi: 10.1213/XAA.0000000000000914. PMID 30844822
- [Background] Holland EL, Bosenberg AT. Early experience with erector spinae plane blocks in children. Paediatr Anaesth. 2020 Feb;30(2):96-107. doi: 10.1111/pan.13804. Epub 2020 Jan 27. PMID 31883421